CLINICAL TRIAL: NCT02885194
Title: Impact of Subthalamic Nucleus Deep Brain Stimulation on Pain in Parkinson Disease : Clinical and Neurophysiological Study
Brief Title: Impact of Subthalamic Nucleus Deep Brain Stimulation on Pain in Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2014.866
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Pain; Deep Brain Stimulation; Laser-Evoked Potentials
MeSH Terms: conditions — Parkinson Disease; Pain | interventions — Laser-Evoked Potentials

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients who underwent Deep Brain Stimulation (DBS) (Other): Patients who underwent Subthalamic Nucleus (STN)-DBS at Lyon
  Interventions: Other: Laser-Evoked potential

INTERVENTIONS:
Other: Laser-Evoked potential — Laser-Evoked potential can document lesions of spinothalamic tract and lateral brainstem and of thalamo-cortical projections conducting nociceptive signals. The rapid heating of skin by infrared laser pulses stimulate small fibers sensory pathways. The main cortical laser evoked potential is a complex of components N2-P2. Evaluation of the registered potentials includes shape, latency and amplitude.

SUMMARY:
Pain is a common symptom of Parkinson's disease (PD) but the physiology remains poorly understood. Recent work suggests that subthalamic nucleus deep brain stimulation (STN-DBS) could make a profit on the pain in PD.

The investigator would drive a study with a follow up of PD patients before and after STN-DBS. The pain will be clinically explored by targeted questionnaires and electrophysiological through laser evoked potentials.

The questionnaires are designed to quantify and characterize the pain in these patients. Laser evoked potentials will, through repetitive stimulation, study both the functional status of the afferent nociceptive pathways, their habituation to repetitive nociceptive stimuli, and so better understand any abnormalities of the central processing of nociceptive information.

ELIGIBILITY:
Inclusion Criteria:

* A patient with idiopathic Parkinson's disease
* Age between 30 and 70 inclusive.
* No cognitive decline (MMS greater than or equal to 24)
* Normal brain MRI
* Informed consent signed
* With or without pain sensation

Exclusion Criteria:

* Presence of other neurological pathology that could explain the pain.
* MMS less than 24
* Pregnant or breastfeeding women

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Modification of habituation in percentage, between tests performed before and after DBS | After the second laser evoked potential which occurred around 3 months after STN-DBS
  The habituation is the change of amplitude between the first and the second response of the double stimulation during the laser evoked potential. We calculated a percentage

SECONDARY OUTCOMES:
Change in latency of laser evoked potential responses before and after DBS | After the second laser evoked potential which occurred around 3 months after STN-DBS
  latency is calculated in millisecond
Change in amplitude of laser evoked potential responses before and after DBS | After the second laser evoked potential which occurred around 3 months after STN-DBS
  amplitude is calculated in microvolts

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane THOBOIS, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Service de Neurologie C, Hôpital Neurologique, HCL, Bron, France

IPD SHARING:
Plan to Share IPD: No